CLINICAL TRIAL: NCT05568186
Title: Correlation Between Different Thermal Patterns of Infrared Thermal Imaging and Clinical Phenotype and Prognosis in Patients With Postherpetic Neuralgia
Brief Title: Correlation Between Thermal Patterns of Infrared Thermal Imaging and Clinical Phenotype in Patients With Postherpetic Neuralgia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xianwei Zhang，MD (Other)
Responsible Party: Sponsor-Investigator, Xianwei Zhang，MD, professor, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Other Study IDs: postherpetic neuralgia
Record Dates: First submitted 2022-10-01; First posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Postherpetic Neuralgia; Infrared Thermal Imaging
Keywords: postherpetic neuralgia; infrared thermal imaging; clinical phenotype; disease course
MeSH Terms: conditions — Neuralgia, Postherpetic; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Postherpetic neuralgia (PHN) is the most frequent complication of herpes zoster(HZ) and is defined as pain persisting for >1month after the healing of herpetic skin lesion or pain persisting for > 3 months following the onset of HZ. PHN manifests as spontaneous throbbing, stabbing, or burning, usually accompanied by various abnormal sensory symptoms , which affect 5-20% of patients with HZ. Due to the lack of accurate and objective auxiliary examination tools, it is difficult for diagnosis and treatment of PHN. As a non-invasive examination method, infrared thermal imaging (IRT) can play a role in the diagnosis and treatment of neuropathic pain by objectively reflecting the changes and distribution characteristics of human body surface temperature. However, there are few studies on the relationship between clinical phenotype and thermal infrared image temperature changes in PHN patients, and the relationship between the thermal pattern of skin temperature and the duration of disease and treatment progress in PHN patients has not been fully elucidated. This study was conducted to investigate the relationship of thermal imaging data with the duration of the disease, clinical phenotype, treatment effect, in order to explore the role of infrared thermal imaging in the diagnosis and treatment of PHN. Methods：all PHN patients will included. At each visit, a pain NRS score was performed, and clinical phenotypes were tested and labeled, including: allodynia, numbness, itching, heat sensation, cold sensation, and the most painful area(MPA). Infrared thermal imaging was performed, the Average Relative Temperature (ART) within the affected area and the contralateral area was compared. The relationship between the temperature change and duration of the disease, clinical phenotype, treatment effect was assessed.

DETAILED DESCRIPTION:
patients with the follow conditions were excluded: 1)The skin area was lesions because of other disease(trauma, inflammation, skin scar, skin disease, tumor, etc.); 2) history of psychiatric diseases, chronic pain. 3) inabilities to complete IRT examination.

ELIGIBILITY:
Inclusion Criteria:

* 1) patients>18 years-old 2) pain lasts at least 1 month after lesion crusting 3) Agreed to participate the research

Exclusion Criteria:

* 1))the skin area was lesions because of other disease(trauma, inflammation, skin scar, skin disease, tumor, etc.); 2) history of psychiatric diseases, chronic pain. 3)inabilities to complete IRT examination. 4) Disagree to participate to the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all PHN patients in our hospital
Sampling Method: Non-Probability Sample
Enrollment: 166 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Thermal pattern difference between affected side and contralateral side | 1 year
  Thermal pattern difference between affected side and contralateral side
temperature difference between affected side and contralateral side | 1 year
  temperature difference between affected side and contralateral side

SECONDARY OUTCOMES:
the relationship between the temperature change and disease duration | 1 year
  the relationship between the temperature change and disease duration
the relationship between the temperature change and Pain Scores on Visual Analog Scale at each visit | 1 year
  the relationship between the temperature change and Pain Scores on Visual Analog Scale at each visit
the relationship between the temperature change and clinical phenotype | 1 year
  the relationship between the temperature change and clinical phenotype
the relationship between the temperature change and treatment effect | 1 year
  the relationship between the temperature change and treatment effect

CONTACTS AND LOCATIONS:
Overall Officials: Xianwei Zhang, Doctor, Principal Investigator — Huazhong University of Science and Technology
Locations (1):
- Department of Anesthesiology, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China